CLINICAL TRIAL: NCT01557829
Title: Clinical Study of the Amedica Corporation Valeo OL Interbody Fusion Devices for Posterior Lumbar Interbody Fusion
Brief Title: Valeo OL Interbody Fusion Devices for Posterior Lumbar Interbody Fusion SNAP Trial
Acronym: SNAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amedica Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Amedica 2011-9; NL34808.100.10 (Registry Identifier: Netherlands Clinical Trials Registry)
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Disc Degeneration of Pfirrmann Grade III or Greater; Degenerative Spondylolisthesis; Isthmic Spondylolisthesis of Grade I or II
Keywords: spondylolisthesis; disc degeneration; lumbar interbody fusion; randomized controlled trial; ceramic interbody spacer
MeSH Terms: conditions — Spondylolisthesis; Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEEK interbody cage (Active Comparator): Posterior fusion with an interbody spacer (cage) made from polyetheretherketone (PEEK) plastic. The open space in the center of the cage is filled with local bone or bone harvested from the iliac crest.
  Interventions: Device: Posterior lumbar interbody fusion with a PEEK cage
- Valeo OL ceramic cage (Experimental): Posterior fusion with the Valeo OL cage, a silicon nitride ceramic interbody spacer. The center area of the cage is filled with autograft local bone or bone harvested from the iliac crest.
  Interventions: Device: Posterior lumbar interbody fusion with a Valeo OL cage

INTERVENTIONS:
Device: Posterior lumbar interbody fusion with a PEEK cage — PEEK cage suitable for oblique placement in the lumbar spine
  Other Names: Amedica Phantom Plus or Pioneer Bullet-Tip cage
  Arms: PEEK interbody cage
Device: Posterior lumbar interbody fusion with a Valeo OL cage — Posterior lumbar interbody fusion with a single Valeo OL ceramic cage.
  Other Names: Valeo OL; silicon nitride ceramic
  Arms: Valeo OL ceramic cage

SUMMARY:
This study randomizes degenerative spondylolisthesis and/or degenerative disc patients into two groups: one to receive a new ceramic implant and a control group with a more traditional PEEK plastic implant. The procedure uses a single oblique cage in each group. The study will measure and compare pain and disability improvement with the two implanted devices over a period of two years. The fusion status will also be judged with plane x-rays and one CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18-75 years
* Chronic low back pain unresponsive to at least six months of conservative care
* MRI and standing x-ray evidence of Pfirrmann Grade III or greater disc degeneration and/or degenerative or isthmic spondylolisthesis of Grade I or II

Exclusion Criteria:

* Osteoporosis
* Patients with prior failed fusion at the same level
* Degenerative scoliosis
* Degenerative spondylolisthesis greater than Grade II
* Pregnancy
* Psychiatric or mental disease
* Alcoholism (drinking more than 5 units per day)
* Active infection or prior infection at the surgical site
* Active cancer
* Insufficient language skills to complete questionnaires
* Participation in another study
* More than two symptomatic levels that need fusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-02; Primary Completion 2016-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire (RMDQ) | 12 months post-op
  The improvement in the RMDQ over the pre-op RMDQ value for each group will be compared

SECONDARY OUTCOMES:
Fusion status | 3 mo., 6 mo., 12 mo., 24 months
  Plane film radiographs will be used to assess fusion at all four follow-up periods. At 12 months a CT scan will be performed.
Oswestry Disability Index (ODI) | 12 months post-op
  The improvement in the ODI over the pre-op ODI for each Group

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Medical Center Haaglanden, The Hague
  - Diakonessenhuis, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kersten RF, van Gaalen SM, Arts MP, Roes KC, de Gast A, Corbin TP, Oner FC. The SNAP trial: a double blind multi-center randomized controlled trial of a silicon nitride versus a PEEK cage in transforaminal lumbar interbody fusion in patients with symptomatic degenerative lumbar disc disorders: study protocol. BMC Musculoskelet Disord. 2014 Feb 25;15:57. doi: 10.1186/1471-2474-15-57. PMID 24568365